CLINICAL TRIAL: NCT06383195
Title: The Reliability and Validity of the Ankylosing Spondylitis Performance Index (ASPI) Physical Function Test in Enthesitis-Related Arthritis
Brief Title: The Reliability and Validity of the Ankylosing Spondylitis Performance Index (ASPI) in Enthesitis-Related Arthritis
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sinan Buran, Principal Investigator, Hacettepe University
Other Study IDs: SBA 24/189
Record Dates: First submitted 2024-04-17; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Enthesitis Related Arthritis; Enthesitis Related Arthritis, Juvenile
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study assesses the test-retest reliability, construct validity, and minimal detectable change of the Ankylosing Spondylitis Performance Index (ASPI) in assessing the physical function of patients with Enthesitis-related arthritis (ERA).

DETAILED DESCRIPTION:
Enthesitis-related arthritis (ERA), which is considered the counterpart of adult spondyloarthropathies, is a human leukocyte antigen (HLA) B27-related subtype of juvenile idiopathic arthritis (JIA) characterized by enthesitis and arthritis, which can also affect the sacroiliac joints and axial spine. Compared to other JIA categories, ERA patients tend to have higher pain intensity, lower physical functionality, and poorer health status. Maintaining or improving physical functionality is one of the primary treatment goals for ERA patients. Physical functionality is also considered an important outcome measure for assessing disease course and effectiveness of treatment. When the literature is examined, it is seen that self-report-based questionnaires are used more frequently, and performance-based measurements are used less in the evaluation of ERA patients.

The Ankylosing Spondylitis Performance Index (ASPI) is a physical performance test that consists of a combination of three reliable tests (bending, putting on socks, and standing up from the floor) developed from the Bath Ankylosing Spondylitis Functional Index (BASFI). It is reported that applying ASPI can provide more objective information about the improvement in physical functionality and a better estimate of the patients' abilities.

ASPI has significant potential in this disease group, considering factors such as the fact that it was developed in adult spondyloarthropathy patients, which is the equivalent of ERA. However, its psychometric properties must be appropriate for the ASPI to be used in clinical settings and research. To our knowledge, no studies have been conducted in the current literature on the validity and reliability of the ASPI in ERA patients. Therefore, this study aimed to evaluate the test-retest reliability, construct validity, and minimal detectable change of the ASPI in assessing the physical function of patients with ERA.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Enthesitis-Related Arthritis (ERA) according to The International League of Associations for Rheumatology (ILAR) classification
* Being between the ages of 7-18
* Volunteering to participate in research

Exclusion Criteria:

* Advanced heart/lung/liver/kidney disease, neurological disease and malignancies
* Having undergone major orthopedic surgery
* The presence of moderate to severe mental problems that will negatively affect participation
* Not volunteering to participate in the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Enthesitis-related arthritis (ERA)
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Ankylosing Spondylitis Performance Index (ASPI) | Baseline (First assessment)
  The ASPI is performed in a common consultation room and consists of 3 standardized performance tasks: (1) bending to pick up 6 pencils from the floor (one by one); (2) putting on socks (mean of 3 times); and (3) getting up from the floor (mean of 3 times). The completion time for each task in the test will be recorded in seconds. The pain the patient feels during each task in the test will be evaluated using the Numeric Rating Scale (NRS) (0: no pain and 10: extreme pain). In addition, the patient's exertion in each task in the test will be evaluated using the Borg scale (0: no exertion and 10: extreme exertion).

SECONDARY OUTCOMES:
Childhood Health Assessment Questionnaire (CHAQ) | Baseline (First assessment)
  The CHAQ assesses the functional abilities of children with JIA in activities of daily living. It comprises eight sections (dressing and grooming, arising, eating, walking, hygiene, reaching, griping, and activities) and evaluates pain (0: no pain and 10: extreme pain) and general well-being (0: no problem and 10: extreme problem) using a Visual Analog Scale. The total CHAQ score ranges from 0 to 3 (higher scores reflect low functionality).
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline (First assessment)
  The BASDAI was used to determine the disease activity levels of the patients. This index consists of 6 items related to 5 symptoms that occurred during the previous week: fatigue, spinal pain, joint pain/swelling, tenderness, and morning stiffness. The total BASDAI score ranges from 0 to 10 (higher scores reflect greater disease activity).
Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline (First assessment)
  The BASFI was used to determine the functional levels of the patients. This index has 10 questions evaluating the daily living activities. The total BASFI score ranges from 0 to 10 (higher scores reflect a greater impairment).
Bath Ankylosing Spondylitis Metrology Index (BASMI) | Baseline (First assessment)
  The BASMI is composed of five measurements: cervical rotation, tragus-to-wall distance, lateral flexion, modified Schober's distance, and intermalleolar distance. Each measurement indicates either 0 (mild disease involvement), 1 (moderate disease involvement), or 2 (severe disease involvement) points, resulting in a total BASMI score of 0-10.
Modified Paediatric Mini Mental Scale (MPMMS) | Baseline (First assessment)
  MPMMS is a scale developed to determine children's cognitive skills and is recommended for use by professionals in various healthcare settings.

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Buran, RA, Principal Investigator — Hacettepe University Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No